CLINICAL TRIAL: NCT01396668
Title: Phase Ⅱ Trial of Fixed Dose Rate Gemcitabine and Cisplatin Chemotherapy Followed by Chemoradiation With Capecitabine in Patients With Locally Advanced Pancreatic Cancer
Brief Title: Fixed Dose Rate Gemcitabine and Cisplatin Followed by Chemoradiation for Locally Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Seock-Ah Im, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-0412-138-005
Record Dates: First submitted 2011-07-01; First posted 2011-07-19 (Estimated); Last update posted 2011-07-19 (Estimated); Status verified 2011-07

CONDITIONS: Pancreatic Cancer
Keywords: locally advanced
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Cisplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: gemcitabine, cisplatin, capecitabine — Gemcitabine: 1000mg/㎡ (day 1, 8), cisplatin 60mg/㎡ (day 1) Capecitabine: 650mg/㎡ twice a day, during radiotherapy Gemcitabine: 1000mg/㎡ (day 1, 8)

SUMMARY:
This is a phase Ⅱ trial of fixed dose rate gemcitabine and cisplatin chemotherapy followed by chemoradiation with capecitabine in patients with locally advanced pancreatic cancer.

DETAILED DESCRIPTION:
The main purpose of this study is to evaluate the efficacy and safety of fixed dose rate gemcitabine and cisplatin chemotherapy followed by chemoradiation with capecitabine in patients with locally advanced pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* unresectable locally advanced pancreatic cancer
* no distant metastasis
* histologically confirmed adenocarcinoma of pancreas
* 18-75 of age
* ECOG performance status 0-2
* normal marrow function :

  * WBC at least 3,000/mm3 OR Absolute neutrophil count at least 1,500/mm3
  * Platelet count at least 100,000/mm3
* normal liver function :

  --Bilirubin no greater than 2.0 mg/dL AST less than 3 times upper limit of normal (ULN)
* normal renal function :

  --Creatinine no greater than 1.5 times ULN
* signed informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2004-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Time to progression | 12 months

SECONDARY OUTCOMES:
safety | 12 months
  number of patients who experienced grade 3-4 toxicity by NCI-CTCAE
1 year survival rate | 1 year
response rate | 1 year
  response rate by RECIST criteria
overall survival | 1 year
clinical benefit rate | 1 year
  CR+PR+SD by RECIST criteria

CONTACTS AND LOCATIONS:
Overall Officials: Seock-Ah Im, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (2):
- South Korea (2):
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul